CLINICAL TRIAL: NCT03750149
Title: Reading Analysis in Ophthalmologic Patients: a Pilot Study
Brief Title: Reading Analysis in Ophthalmologic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TRC
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Maculopathy; Age Related Macular Degeneration; Glaucoma; Epiretinal Membrane
Keywords: Diabetic Maculopathy; Age Related Macular Degeneration; Glaucoma; Epiretinal membrane; Reading analysis
MeSH Terms: conditions — Macular Degeneration; Glaucoma; Epiretinal Membrane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ophthalmologic Disease (Experimental): Patients with glaucoma, AMD, diabetic maculopathy, epiretinal membranes, and healthy patients will undergo a reading analysis using the EyeTracker
  Interventions: Device: EyeTracker

INTERVENTIONS:
Device: EyeTracker — Patients with various ophthalmologic diseases (ERM, glaucoma, AMD, diabetic retinopathy) will undergo reading analysis using the EyeTracker

SUMMARY:
Investigation of the reading parameters and fixation behavior in patients with different ocular diseases (age-related macular degeneration, glaucoma, diabetic maculopathy, epiretinal membrane) and healthy subjects. In addition, fixation analysis and retinal sensitivity measurements will be done with a microperimeter in each subject.

DETAILED DESCRIPTION:
Reading is a complex function. It requires a proper retinal image that is received by the brain. There it is analyzed for letter and word recognition and then the semantics is detected. Reading speed slows down when letters are blurred, or do not have enough contrast or luminance or when binocular fusion is hampered. Hence, it is obvious that reading ability is reduced in patients with various ocular diseases. Especially, pathologies effecting the posterior pole (central and paracentral vision) might impair reading parameters significantly.

Recently, the Eyetracker Eyelink 1000 (SR Research Ltd, Canada) became available. It´s application was described previously. Briefly, a high-speed infrared camera detects the position of eye (pupil and corneal reflex) and in turn the direction of gaze 500 times per second. During the calibration process the position can be linked to the position on a screen where, for instance, a text or a fixation target can be projected. Direction of gaze is recorded during the reading process and the gathered data are analyzed.

Fixation ability was assessed using Eyelink 1000 in patients with age-related macular degeneration. It was shown that fixation is related to visual function. The worse eye showed reduced fixation ability which is improved during binocular fixation. This study investigates reading parameters in patients with various ocular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Absence of ocular disease (Group 1)
* Present ocular disease (age-related macular degeneration, glaucoma, diabetic maculopathy, epiretinal membrane/macular hole) as judged by the investigator (Group 2 - 5)
* Maximum of allowed cylinder-power in the spectacles: +1.50D

Exclusion Criteria:

* Ocular pathologies, that may interfere with study measurements, such as corneal scars
* In case of pregnancy (pregnancy test will be taken prior to inclusion into the study in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Reading speed | 12 months
  Reading speed (words per minute) will be analysed using the EyeTracker device. The patient has to read 4 texts with different contrast levels. The faster the patient can read a text, the better the results.

SECONDARY OUTCOMES:
Retinal perimetry | 12 months
  Analysis of retinal fixation will be done using microperimetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided